CLINICAL TRIAL: NCT00259025
Title: The Effect of Intravenous n-3 Polyunsaturated Fatty Acids on Risk Markers for Sudden Cardiac Death in Hemodialysis Patients
Brief Title: Intravenous n-3 Fatty Acids and Sudden Cardiac Death in Hemodialysis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IVN3DIALYSE
Record Dates: First submitted 2005-11-25; First posted 2005-11-29 (Estimated); Last update posted 2008-08-11 (Estimated); Status verified 2008-04

CONDITIONS: Renal Failure, Chronic
Keywords: Renal failure, chronic; Death, sudden, cardiac; Heart rate variability; Tachycardia, ventricular; Ventricular premature complexes; Ventricular repolarization; Eicosapentaenoic acid; Docosahexaenoic acid
MeSH Terms: conditions — Kidney Failure, Chronic; Death, Sudden, Cardiac; Tachycardia, Ventricular; Ventricular Premature Complexes

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Drug: lipid emulsion with a high content of n-3 fatty acids

SUMMARY:
The main purpose of this study is to investigate whether intravenous infusion of a lipid emulsion with a high content of n-3 polyunsaturated fatty acids can improve heart rate variability and ventricular repolarization and reduce ventricular arrhythmias in hemodialysis patients.

DETAILED DESCRIPTION:
Cardiovascular disease is the most common cause of death in haemodialysis (HD)patients, and half of these deaths are due to sudden cardiac death caused by ventricular arrhythmias. HD patients have an attenuated heart rate variability (HRV) and a high frequency of ventricular arrhythmias, both of which are predictors of sudden cardiac death(SCD). n-3 polyunsaturated fatty acids (PUFA) improves HRV and reduces the risk of SCD. n-3 PUFAs are obtained from fatty fish and fish oil and are incorporated into cell membranes after long-term ingestion. However, it is not known if this incorporation is essential or merely serves as storage for n-3 free PUFAs to be release during for instance myocardial ischaemia.

The study hypothesis is that intravenous infusion of a lipid emulsion with a high content of n-3 PUFAs will improve HRV and ventricular repolarization and reduce ventricular arrhythmias via an acute increase in free non-esterified n-3 PUFAs in plasma.

In a randomized, placebo-controlled design a n-3 PUFA rich emulsion (or placebo) will be administered during hemodialysis treatment. The two study groups will be compared with respect to heart rate variability, ventricular repolarization parameters, ventricular ectopic beats and arrhythmias and the content of n-3 PUFA in plasma and cell membranes will be compared.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 yrs
* End-stage renal failure
* Maintenance haemodialysis treatment > 3 months

Exclusion Criteria:

* Allergy to fish or egg protein
* Body weight < 50 kgs
* Chronic supraventricular tachycardia
* Implanted pacemaker
* Myocardial infarction within 6 months
* PCI or CABG within 6 months
* Stroke or TIA within 6 months
* HbA1C > 10 %
* ALAT > 100 U/l
* Triglycerides > 3 mmol/l
* Ongoing infection
* Tendency to severe blood pressure drops during dialysis treatment
* Malignancy
* Psychiatric disorder
* Pregnancy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-09; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Heart rate variability

SECONDARY OUTCOMES:
Ventricular repolarization, ventricular arrhythmias
n-3 polyunsaturated fatty acids in plasma and cell membranes

CONTACTS AND LOCATIONS:
Overall Officials: Jeppe H Christensen, MD, DMSci, Principal Investigator — Aalborg Sygehus
Locations (1):
- Department of Nephrology, Aalborg Hospital, Aalborg, Denmark